CLINICAL TRIAL: NCT04085744
Title: A Comparison Between Local Anesthetics and Topical Cortikosteroids That is Applied to the Area of Cuff of Tracheal Intubation Tube in Pediatric Patients
Brief Title: A Comparison Of Local Anesthetic Agents And Steroid On Tracheal Tube Cuff
Acronym: LA-STEROID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ALI ULVI OLC, Principal Investigator, Derince Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AOLC-1
Record Dates: First submitted 2019-09-07; First posted 2019-09-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia Intubation Complication; Intubation Complication; Sore Throat
Keywords: intubation; anesthesia; corticosteroids; lidocaine; complication of intubation
MeSH Terms: conditions — Pharyngitis | interventions — Lidocaine; Steroids

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (No Intervention): In this group any drug will be applied on the cuff of the intubation tube
- lidocaine group (Active Comparator): 10% lidocaine spray will be applied on the cuff of the intubation tube topically and patient will be intubated.
  Interventions: Drug: Lidocaine 10% Spray
- steroid group (Active Comparator): mometasone furoate spray will be applied on the cuff of the intubation tube topically and patient will be intubated.
  Interventions: Drug: Mometasone nasal spray

INTERVENTIONS:
Drug: Lidocaine 10% Spray — lidocaine will be apply on the cuff
  Other Names: lidocaine
  Arms: lidocaine group
Drug: Mometasone nasal spray — mometasone spray will be applied on the cuff
  Other Names: steroid
  Arms: steroid group

SUMMARY:
This study aims to compare effects of two different agents on complications due to tracheal tube cuff in pediatric patients. Sore throat, hoarseness, laryngospasm, bronchospasm are the main complications.

DETAILED DESCRIPTION:
In the literature there were studies about both local anesthetic agents and topical steroids and different densities of saline which were applied to decrease airway complications. In this study researchers intended to compare effects of local anesthetic agents and topical steroids applying around tracheal tube on airway complications which may occur in the first 24 hours after surgery. All pediatric patients scheduled for elective surgery will be recruited. enrolled patients will randomly assigned in to three groups: Control group, local anesthetic group and topical steroid group.

ELIGIBILITY:
Inclusion Criteria:

* Being ages between 2 and 18
* undergoing elective surgery
* intubated patients over 1 hour
* ASA(American Society of Anesthesiologists) Class I-II patients

Exclusion Criteria:

* Urgent surgeries
* Tonsillectomies, adenoidectomies ..etc, operations that causes sore throat due to the operation area.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) for pain | 1 hour
  Self Reported VAS at postoperative unit. VAS 0 is no pain VAS 10 is pain as bad as can be
Visual analog scale (VAS) for pain | 6 hours
  Self reported VAS postoperative at hour 6. VAS 0 is no pain VAS 10 is pain as bad as can be
Visual analog scale (VAS) for pain | 12 hours
  Self reported VAS postoperative at hour 12. VAS 0 is no pain VAS 10 is pain as bad as can be
Visual analog scale (VAS) for pain | 24 hours
  Self reported VAS at postoperative hour 24. VAS 0 is no pain VAS 10 is pain as bad as can be

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Z Turan, Study Director — HEALTH AND SCİENCE UNIVERSITY DERINCE TRAINING AND RESEARCH HOSPITAL
Locations (1):
- Health and Science University Derince Training and Research Hospital, Derince, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No